CLINICAL TRIAL: NCT06530459
Title: The MUScle Strengthening Exercises and Estrogen (MUSE) Randomized Controlled Trial for Menopausal Arthralgia
Brief Title: The MUSE Study for Menopausal Arthralgia
Acronym: MUSE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Professor, National University Hospital, Singapore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00727
Record Dates: First submitted 2024-04-11; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Arthralgia; Menopause; Perimenopausal Disorder; Joint Pain; Postmenopausal Disorder
Keywords: Menopausal hormone therapy; Muscle strength; Exercise; Randomized controlled trial; Midlife women
MeSH Terms: conditions — Arthralgia; Motor Activity | interventions — Hormone Replacement Therapy; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise (Experimental): Curated exercises designed to address specific muscle groups and joints that are painful and problematic.
  Exercises would focus on upper and lower body strength generally. It is anticipated that participants ideally should exercise at least 3 times per week based on the strength training prescription. They could potentially exercise everyday, alternating between upper and lower body strength training.
  Interventions: Behavioral: Exercise training
- Menopausal hormone therapy (Experimental): Menopausal hormone therapy comprising: 17beta-estradiol topical gel (1.25-2.5 gms) applied daily, and micronized Progesterone 200mg daily for 12 days each month.
  Interventions: Drug: Menopausal hormone therapy
- Combination of exercise and menopausal hormone therapy (Experimental): 1. Curated exercises designed to address specific muscle groups and joints that are painful and problematic.
     Exercises would focus on upper and lower body strength generally. It is anticipated that the participants ideally should exercise at least 3 times per week based on the strength training prescription. They could potentially exercise everyday, alternating between upper and lower body strength training.
  2. Menopausal hormone therapy comprising: 17beta-estradiol topical gel (1.25-2.5 gms) applied daily, and micronized Progesterone 200mg daily for 12 days each month.
  Interventions: Combination Product: Menopausal hormone therapy + exercise training
- Standard care (No Intervention): Standard care will be provided.

INTERVENTIONS:
Drug: Menopausal hormone therapy — Apply 17 beta-Estradiol topical gel (1.25-2.5 gms) daily Ingest Micronized Progesterone 200mg daily for 12 days each month
  Arms: Menopausal hormone therapy
Behavioral: Exercise training — Exercises would focus on upper and lower body strength generally. It is anticipated that the participants ideally should exercise at least 3 times per week based on the strength training prescription. They could potentially exercise everyday, alternating between upper and lower body strength training. In all, there are up to 1-2 in-person therapy sessions and home sessions at least 3 times per week.
  Arms: Exercise
Combination Product: Menopausal hormone therapy + exercise training — 1. Apply 17 beta-Estradiol topical gel (1.25-2.5 gms) daily and Ingest Micronized Progesterone 200mg daily for 12 days each month
  2. Exercises would focus on upper and lower body strength generally. It is anticipated that patients ideally should exercise at least 3 times per week based on the strength training prescription. They could potentially exercise everyday, alternating between upper and lower body strength training. In all, there are up to 1-2 in-person therapy sessions and home sessions at least 3 times per week.
  Arms: Combination of exercise and menopausal hormone therapy

SUMMARY:
The investigators plan to conduct a pilot 4-arm, randomized study comprising the following interventions: muscle strengthening exercises (MSE) alone, estrogen therapy (ET) alone, and a combination of MSE and ET, compared to usual care in women with menopausal arthralgia. The aim of this pilot study is to assess the feasibility, patient acceptability, and patient perspectives and logistics of delivering interventions, and practicability of outcome assessment tools in this 4-arm study over a 12-week period.

DETAILED DESCRIPTION:
Recruited participants will be randomized to one of the following arms for 12 weeks: usual clinical care, 17b-Estradiol/progesterone (ET) only, Muscle strengthening exercises (MSE) only, combination of MSE plus ET. All participants will be assessed at Baseline and at 12 weeks.

Estrogen therapy (ET): Participants would apply 17b-estradiol (1.25-2.5 gms/daily) gel transdermally to joints and muscles most affected by arthralgia for 12 weeks. Participants with intact uteri would also be issued micronized Progesterone 200mg tablets to be taken orally for 12 days each month. Medications would be dispensed by the National University Hospital (NUH) pharmacy.

Muscle strengthening exercises (MSE) Exercises would be demonstrated in person by qualified staff physiotherapists. All Participants would be given a standard strength training protocol, with additional tailored exercises targeting their pain conditions, abilities and personal preferences. Exercises would focus on upper and lower body strength generally. Participants would be encouraged to exercise every day, alternating between upper and lower body strength training following the curated exercises. Exercise regimes would be reinforced through weekly reminders, and posts through social media.

MSE plus ET: Participants randomized to combination of would have both treatments administered at the same time within the same intervention period of 12 weeks. In other words, participants would be instructed to do the curated exercises and apply 17b-estradiol (1.25-2.5 gms/daily) gel trans-dermally with micronized progesterone oral tablets.

Usual care: Participants would continue their usual daily routines and come for outcome assessments at baseline and 12 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with muscle stiffness and joint discomfort in various sites, including hands, knees, back, hips, and/or shoulders. Patients with pain in only one isolated joint would not be accepted.
2. Arthralgia symptoms with onset, or has become worse, over the perimenopausal or early postmenopausal period (within 5 years of the menopause).
3. Women should be at the menopause transition, less than or equal to 59 years old at the time of enrollment, or within 5 years of menopause whichever is earlier.

   .
4. Arthralgia for at least 3 months (pain lasting beyond normal injury healing period)
5. Community-dwelling and able to ambulate independently.

EXCLUSION CRITERIA:

1. History of thrombo-embolic diseases, strokes, ischemic heart disease, dementia or psychiatric disorders, active liver disease or renal impairment, severe hyperlipidemia, gout, thyroid disease, systemic lupus erythematosus, rheumatoid arthritis, or other chronic inflammatory conditions.
2. Pregnancy
3. Non-adherence to national guidelines for breast cancer screening
4. High risk for breast cancer
5. Any joint surgery within the last 6 months
6. Severe obesity: BMI>35
7. Migraine with aura
8. Poorly controlled diabetes
9. Use of any form of female hormone supplementation within the past 12 weeks.
10. High venous thromboembolism risk
11. Current cholecystitis, fibroids, or undiagnosed abnormal uterine bleeding.
12. Current smoker.
13. History of endometrial, ovarian, peritoneal, cervical, breast or endocrine-dependent cancers.
14. Receiving treatment for any form of cancer.
15. History of fragility bone fractures within the 2 years.
16. Any other cognitive, musculoskeletal, neurological, and cardiorespiratory condition affecting one's ability to participate in the study.

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Relative changes in perceived arthralgia at the end of intervention | After 12 weeks of intervention
  Relative changes in perceived arthralgia with the 10-item Örebro Musculoskeletal Pain Screening Questionnaire (Short Form) would be the pre-specified primary outcome parameter.
  Participants would be asked to rank each item on a 11-point scale from 0 to 10.

SECONDARY OUTCOMES:
Changes in Handgrip strength (kg) | After 12 weeks of intervention
  Handgrip strength (kg) will be assessed twice on each arm, using the Jamar dynamometer.
Changes in isokinetic knee extension strength (degree/second) | After 12 weeks of intervention
  The knee extension strength test will be conducted using the isokinetic dynamometry with Biodex, and measured in degree/second.
Changes in physical performance using the Physical Performance Battery | After 12 weeks of intervention
  The investigators will use a modified version of the lower-extremity performance tests conducted in the Established Populations for the Epidemiologic Studies of the Elderly, wherein scores from four tests will be added to form a continuous score ranging from 0 to 4.
Changes in associated menopausal symptoms using the Menopause Rating Scale (MRS) | After 12 weeks of intervention
  Menopausal symptoms will be assessed using the Menopause Rating Scale (MRS), comprising 11 menopausal symptoms. Each symptom will be scored from 0-4 (none, mild, moderate, severe, and extremely severe).
Changes in sleep quality using the Pittsburgh Sleep Quality Index (PSQI) | After 12 weeks of intervention
  The Pittsburgh Sleep Quality Index will be used to assess perceived sleep habits in the past month, with a maximum score of 21 points.
Changes in anxiety symptoms using the GAD-7 | After 12 weeks of intervention
  Anxiety symptoms will be assessed by the General Anxiety Disorder Scale (GAD-7), and scoring ranges from 0 to 21 points.
Changes in depression symptoms using the CES-D | After 12 weeks of intervention
  Depressive symptoms will be assessed using the Center for Epidemiologic Studies for Depression Scale (CES-D). The maximum score is 60.
Changes in perceived quality of life using the SF-12. | After 12 weeks of intervention
  The 12-Item Short Form Survey (SF-12) will be used to assess quality of life.
Changes in verbal memory measured using the Hopkins Verbal Learning Test | After 12 weeks of intervention
  The Hopkins Verbal Learning Test will be used to assess delays in recall and retention of 12 words.
Changes in insulin resistance using HOMA-IR | After 12 weeks of intervention
  Fasting blood glucose and insulin will be measured to obtain the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No